CLINICAL TRIAL: NCT02945826
Title: uPAR-PET/MRI in Glioblastoma Multiforme
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dorthe Skovgaard, Principal investigator, MD, Phd, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK2016-2; 2016-002417-21 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma Multiforme
Keywords: urokinase plasminogen activator receptor; positron emission tomography; glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- uPAR PET/MRI (Experimental): One injection of 68Ga-NOTA-AE105 followed by PET/MRI.
  Interventions: Drug: One injection of 68Ga-NOTA-AE105; Device: PET/MRI

INTERVENTIONS:
Drug: One injection of 68Ga-NOTA-AE105 — One injection of 68Ga-NOTA-AE105
Device: PET/MRI — Following injection of 68Ga-NOTA-AE105 the patients will be subjected to PET/MRI of the brain

SUMMARY:
The purpose of this study is to investigate the applicability of urokinase plasminogen activator receptor (uPAR) Positron Emission Tomography (PET) / MRI molecular imaging of glioblastoma.

DETAILED DESCRIPTION:
68Ga-NOTA-AE105 is a radioligand targeting urokinase plasminogen activator receptor (uPAR), which is a promising imaging biomarker of tumor aggressiveness. 68Ga-NOTA-AE105 PET/MRI will be applied in patients suspected of glioblastoma multiforme. The uptake of the radioligand 68Ga-NOTA-AE105 will be compared and correlated with expression of the molecular target: uPAR using immunohistochemistry of tumor tissue samples obtained during routine stereotactic biopsies or operation. In addition, the semiquantitative uptake (standard uptake values, SUVs) of 68Ga-NOTA-AE105 in tumor tissue will be correlated with overall survival and progression free survival

ELIGIBILITY:
Inclusion Criteria:

* Patients where imaging with MRI or CT is suspicious of having glioblastoma multiforme, and patients, and who is referred for stereotactic biopsy, chemotherapy or surgery
* The participants must be capable of understanding and giving full informed written consent
* age above 18 years

Exclusion Criteria:

* Pregnancy
* Lactation/breast feeding
* Age above 85 years old
* Weight above 140 kg
* Known allergy towards 68Ga-NOTA-AE105

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
uPAR PET/MRI imaging of uPAR expression | 1 hour
  Standard uptake values (SUVs) of 68Ga-NOTA-AE105 evaluated on uPAR-PET/MRI scan performed within 1 hour following injection of 68Ga-NOTA-AE105, compared with immunohistochemistry of uPAR (semiquantitative)
uPAR PET/MRI prognostic factor for overall survival | 36 months
  Patients will be followed for 36 months after uPAR/PET MRI

SECONDARY OUTCOMES:
uPAR PET/MRI prognostic factor for progression free survival | 36 months
  Patients will be followed for 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Skovgaard, Md, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azam A, Kurbegovic S, Carlsen EA, Andersen TL, Larsen VA, Law I, Skjoth-Rasmussen J, Kjaer A. Prospective phase II trial of [68Ga]Ga-NOTA-AE105 uPAR-PET/MRI in patients with primary gliomas: Prognostic value and Implications for uPAR-targeted Radionuclide Therapy. EJNMMI Res. 2024 Oct 29;14(1):100. doi: 10.1186/s13550-024-01164-9. PMID 39472354